CLINICAL TRIAL: NCT07253246
Title: A Two-Part, Single Ascending Dose and Positron Emission Tomography Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Receptor Occupancy After Single Oral Dose Administration of ENX-205 in Healthy Adult Participants
Brief Title: ENX-205 SAD/PET Study in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Engrail Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ENX-205-001
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 2 of this study is open-label, and as such, randomization and blinding are not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENX-205 (Experimental)
  Interventions: Drug: ENX-205
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENX-205 — oral solution
  Arms: ENX-205
Drug: Placebo — oral solution
  Arms: Placebo

SUMMARY:
This is a two-part study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and receptor occupancy (RO) of ENX-205 in healthy adult participants in a double-blind placebo-controlled, single ascending dose (SAD) study (Part 1) and an open-label, single-dose, positron emission tomography (PET) study (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Biologically female participants who are not pregnant, lactating, or breastfeeding

  1. Of non-childbearing potential, defined as either permanently sterilized, and with a negative pregnancy test. OR
  2. Part 1 only: Of childbearing potential and willing to comply with restrictions related to birth control, and with a negative pregnancy test.
* Biologically male participants (defined as assigned male at birth), if fertile must be willing to comply with restrictions related to birth control. Moreover, male participants should refrain from sperm donation.

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the study or, in the opinion of the Investigator or Sponsor, should not participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Treatment Emergent Adverse events | From Day 1 up to Day 10

SECONDARY OUTCOMES:
Part 2: Number of Participants with Treatment Emergent Adverse events | From Day 1 up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: David George Steel, MBChB, Principal Investigator — Parexel
Locations (1):
- Parexel London EPCU, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No